CLINICAL TRIAL: NCT01957917
Title: Comparing Food and Cash Assistance for HIV-Positive Men and Women on Antiretroviral Therapy in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Ministry of Health and Social Welfare, Tanzania (Other Government)
Responsible Party: Principal Investigator, Sandra McCoy, Assistant Adjunct Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5K01MH094246 (NIH); 5K01MH094246 (NIH)
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: HIV
Keywords: HIV; Food Insecurity; Antiretroviral Therapy
MeSH Terms: interventions — Nutrition Assessment; Counseling; Food Assistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NAC + Food Assistance (Experimental): Arm 1 participants will receive NAC (nutritional assessment and counseling), plus a food ration once a month for 6 months if they continue their regular HIV care.
  Interventions: Other: NAC (Nutritional Assessment and Counseling); Other: Food Assistance
- NAC + Cash Transfer (Experimental): Arm 2 participants will receive NAC (nutritional assessment and counseling), plus a cash transfer equivalent in value to the food transfer once a month for 6 months if they continue their regular HIV care.
  Interventions: Other: NAC (Nutritional Assessment and Counseling); Other: Cash Transfer
- NAC Only (Active Comparator): Arm 3 participants will receive NAC (nutrition assessment and counseling) only, which is the standard of care at the selected health facilities.
  Interventions: Other: NAC (Nutritional Assessment and Counseling)

INTERVENTIONS:
Other: NAC (Nutritional Assessment and Counseling)
Other: Cash Transfer
  Arms: NAC + Cash Transfer
Other: Food Assistance
  Arms: NAC + Food Assistance

SUMMARY:
The importance of good nutrition and food security among people living with HIV infection (PLHIV) is widely recognized. In resource-constrained settings, food insecurity is increasingly recognized as an important barrier to retention in care and adherence to antiretroviral therapy (ART). However, there are few studies demonstrating that food and nutrition assistance programs can improve HIV-related outcomes. This study will address this gap by comparing the effectiveness of three models for short-term support for PLHIV. Food insecure women and men on ART will be randomized into one of three groups: 1) nutrition assessment and counseling (NAC) alone, 2) NAC plus food assistance, or 3) NAC plus cash transfers. The investigators will compare the effect of the three approaches on ART adherence and retention in care after 6, 12, and 24-36 months of follow-up. The investigators hypothesize that NAC plus short-term support in the form of food or cash assistance will result in better adherence to ART and retention in care than NAC alone, and that the effects of NAC plus food assistance will be the same as NAC plus cash assistance. The results from the study will provide evidence about which assistance modalities for PLHIV work best to improve ART adherence and retention in care, and under what conditions. This study will be conducted in Shinyanga Region, Tanzania, where approximately 17 percent of households have poor or borderline food consumption and 7.4 percent of people are living with HIV infection.

DETAILED DESCRIPTION:
The investigators will randomize 785 food insecure women and men who recently initiated ART (determined with the Household Hunger Scale1) into one of three groups: 1) NAC alone , 2) NAC plus food assistance, or 3) NAC plus cash transfers. Food assistance will be a standard food ration consisting of maize flour, groundnuts, and beans. The cash transfer will be the equivalent value as the food ration (approximately $13 USD/month). Participants will receive the monthly food ration or cash transfer for up to six months if they continue to receive monthly HIV care (the standard of care). The investigators will compare the effect of NAC and food or cash assistance to the effect of NAC alone on ART adherence and retention in care at 6, 12, and 24-36 months (Objective #1). The investigators will also compare the effectiveness of NAC plus food assistance and NAC plus cash transfers to determine if their effects are the same (Objective #2).

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age;
2. living with HIV infection;
3. initiated antiretroviral therapy (ART) for HIV infection in the last 90 days;
4. food insecure, as measured with the Household Hunger Scale; and
5. willing and able to provide written informed consent for the study.

Exclusion Criteria:

PLHIV who are severely malnourished (BMI<18.5) will be excluded from the study, as these individuals require therapeutic food support (ready-to-use food products for nutritional recovery). In this study, we will enroll food insecure PLHIV who are at risk of malnutrition but are not severely malnourished (BMI>18.5).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Medication Possession Ratio (MPR) at 6 months and at 12 months | Baseline, 6 months, 12 months
  ART adherence will be measured with the medication possession ratio (MPR), the proportion of time an individual is in possession of >1 ARV or prescription for ARV. MPR is computed as the number of days ARVs are prescribed or dispensed divided by the number of days in the interval, and has been shown to be associated with short-term virologic outcomes. We will determine the proportion of patients with MPR ≥95% in each of the study arms.

SECONDARY OUTCOMES:
Change from baseline in Food Security at 6 months and 12 months | Baseline, 6 months, 12 months
  Food security will be measured with several validated scales: the Household Food Insecurity Access Scale (HFIAS), the Household Hunger Scale (HHS) and the Individual Dietary Diversity Scale (IDDS).
Change from baseline in Viral Suppression at 6 months and 12 months | Baseline, 6 months, 12 months
  viral load <400 copies/mL
Change from baseline in ART adherence at 6 months, 12 months, and 24-36 months | Baseline, 6 months, 12 months, and 24-36 months
  Proportion of patients who report taking at least 95% of prescribed doses in the previous month time frame. This will be measured by self-report.
Change from baseline in Body Mass Index (BMI) at 6 months and 12 months | Baseline, 6, and 12 months
  body weight in kilograms (kg) divided by height in meters squared
Change from baseline in Weight at 6 months and 12 months | Baseline, 6 months, 12 months
Change from baseline of Medication Possession Ratio (MPR) at 12-36 months | 12-36 months
  ART adherence will be measured with the medication possession ratio (MPR), the proportion of time an individual is in possession of >1 ARV or prescription for ARV. MPR is computed as the number of days ARVs are prescribed or dispensed divided by the number of days in the interval, and has been shown to be associated with short-term virologic outcomes. We will determine the proportion of patients with MPR ≥95% in each arm.
Retention in Care at 12-36 months | 12-36 months
  Retention in care will be assessed by number of participants in each arm that are still still in care at 12-36 months

OTHER OUTCOMES:
Change from baseline in ability to work/participation in the labor force at 6 months and 12 months | Baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra I McCoy, PhD, Principal Investigator — University of California, Berkeley
Locations (4):
- Tanzania (4):
  - Kahama District Hospital, Shinyanga, Shinyanga
  - Kambarage Health Center, Shinyanga, Shinyanga
  - Kishapu Health Center, Shinyanga, Shinyanga
  - Shinyanga Regional Hospital, Shinyanga, Shinyanga

REFERENCES:
- [Background] Deitchler M, Ballard T, Swindale A, Coates J. Introducing a Simple Measure of Household Hunger for Cross-Cultural Use. Washington, D.C.: Food and Nutrition Technical Assistance II Project, AED;2011.
- [Background] McMahon JH, Jordan MR, Kelley K, Bertagnolio S, Hong SY, Wanke CA, Lewin SR, Elliott JH. Pharmacy adherence measures to assess adherence to antiretroviral therapy: review of the literature and implications for treatment monitoring. Clin Infect Dis. 2011 Feb 15;52(4):493-506. doi: 10.1093/cid/ciq167. Epub 2011 Jan 18. PMID 21245156
- [Background] Messou E, Chaix ML, Gabillard D, Minga A, Losina E, Yapo V, Kouakou M, Danel C, Sloan C, Rouzioux C, Freedberg KA, Anglaret X. Association between medication possession ratio, virologic failure and drug resistance in HIV-1-infected adults on antiretroviral therapy in Cote d'Ivoire. J Acquir Immune Defic Syndr. 2011 Apr;56(4):356-64. doi: 10.1097/QAI.0b013e3182084b5a. PMID 21191309
- [Background] Goldman JD, Cantrell RA, Mulenga LB, Tambatamba BC, Reid SE, Levy JW, Limbada M, Taylor A, Saag MS, Vermund SH, Stringer JS, Chi BH. Simple adherence assessments to predict virologic failure among HIV-infected adults with discordant immunologic and clinical responses to antiretroviral therapy. AIDS Res Hum Retroviruses. 2008 Aug;24(8):1031-5. doi: 10.1089/aid.2008.0035. PMID 18724803
- [Background] Hong S, Nachega J, Jerger L, et al. Medication Possession Ratio Predictive of Short-term Virologic and Immunologic Response in Individuals Initiating ART: Namibia. 19th Conference on Retroviruses and Opportunistic Infections. Seattle 2012.
- [Background] Coates J, Swindale A, Bilinsky P. Household Food Insecurity Access Scale (HFIAS) for Measurement of Food Access: Indicator Guide. Washington, D.C.: United States Agency for International Development;2007.
- [Background] Swindale A, Bilinsky P. Household Dietary Diversity Score (HDDS) for Measurement of Household Food Access: Indicator Guide (v.2). Washington, D.C.: Food and Nutrition Technical Assistance Project, Academy for Educational Development;2006.
- [Derived] Fahey CA, Njau PF, Kelly NK, Mfaume RS, Bradshaw PT, Dow WH, McCoy SI. Durability of effects from short-term economic incentives for clinic attendance among HIV positive adults in Tanzania: long-term follow-up of a randomised controlled trial. BMJ Glob Health. 2021 Dec;6(12):e007248. doi: 10.1136/bmjgh-2021-007248. PMID 34952856
- [Derived] McCoy SI, Njau PF, Fahey C, Kapologwe N, Kadiyala S, Jewell NP, Dow WH, Padian NS. Cash vs. food assistance to improve adherence to antiretroviral therapy among HIV-infected adults in Tanzania. AIDS. 2017 Mar 27;31(6):815-825. doi: 10.1097/QAD.0000000000001406. PMID 28107221
- [Derived] McCoy SI, Njau PF, Czaicki NL, Kadiyala S, Jewell NP, Dow WH, Padian NS. Rationale and design of a randomized study of short-term food and cash assistance to improve adherence to antiretroviral therapy among food insecure HIV-infected adults in Tanzania. BMC Infect Dis. 2015 Oct 28;15:490. doi: 10.1186/s12879-015-1186-3. PMID 26520572